CLINICAL TRIAL: NCT02997319
Title: Shift Work, Heredity, Insulin, and Food Timing (SHIFT) Study
Brief Title: Shift Work, Heredity, Insulin, and Food Timing Study
Acronym: SHIFT
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Broad Institute of MIT and Harvard (Other); Brigham and Women's Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Richa Saxena, Assistant Professor of Anaesthesia, Massachusetts General Hospital
Other Study IDs: 2016P000651; R01DK105072 (NIH)
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Shift Work Type Circadian Rhythm Sleep Disorder; Diabetes Mellitus, Type 2; Circadian Rhythm Sleep Disorder, Shift Work Type; Insulin Resistance
Keywords: Diabetes Mellitus, Type 2; Insulin Resistance; Shift Work; Circadian Rhythms; MTNR1B
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Disorders, Circadian Rhythm; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, serum insulin, serum glucose, plasma melatonin, blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Night Shift-Workers
- Day Workers

SUMMARY:
The purpose of this study is to determine whether night time eating that coincides with elevated endogenous melatonin impairs glucose tolerance, particularly in carriers of the MTNR1B risk allele.

DETAILED DESCRIPTION:
Preliminary observations suggest that food intake coincident with high melatonin levels leads to impaired glucose tolerance-particularly in MTNR1B risk allele carriers. Our objectives are to determine the effect of concurrent food intake and melatonin on glucose tolerance; and to assess the role of MTNR1B single nucleotide polymorphism (SNP)*melatonin interaction in this deleterious effect. Our central hypothesis is that concurrent high melatonin levels and food intake, commonly experienced in night shift workers, cause long-term impairment of glucose tolerance and that this effect is worse in carriers of the MTNR1B type 2 diabetes (T2D) risk SNP than in non-carriers. The results of this proposal will help to clarify an ongoing controversy about the role of melatonin in glucose tolerance, and will help to develop novel strategies in the prevention and treatment of T2D, especially in shift workers, night eaters, and MTNR1B risk allele carriers.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female
* 18-60 years
* Currently employed (night shift workers and day workers), graduate students, part-time workers, or unemployed
* Able and willing to give consent relevant to genetic investigation

Exclusion Criteria:

* Currently taking any medications for the treatment of diabetes
* Currently taking medications known to affect glycemic parameters, such as glucocorticoids, growth hormone or fluoroquinolones
* Pregnant, nursing or at risk of becoming pregnant
* Chronic renal failure, hepatic diseases, or cancer diagnoses
* Bulimia diagnosis, prone to binge eating
* Eating disorder diagnosis such as anorexia, binge eating, or bulimia
* With psychiatric illness, such as schizophrenia or bipolar affective disorder
* Blind
* History of bariatric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects residing in New England (USA) region
Sampling Method: Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) glucose | Between 0-120 minutes, Visit 2 and 3
  Investigators will measure insulin and glucose levels for 120 minutes at day time and night time visits, and compare them by genotype at selected loci.
Disposition index | Between 0-120 minutes, Visit 2 and 3
  Disposition index will be determined by frequently sampled oral glucose tolerance test

SECONDARY OUTCOMES:
Corrected Insulin Response | Between 0-120 minutes, Visit 2 and 3
Insulin Sensitivity Index | Between 0-120 minutes, Visit 2 and 3
Fasting Glucose | Between 0-120 minutes, Visit 2 and 3
Fasting Insulin | Between 0-120 minutes, Visit 2 and 3
Plasma Melatonin | Between 0-120 minutes, Visit 2 and 3

OTHER OUTCOMES:
Sleep Duration | Total of 2 weeks between Visit 1 and 3
  Sleep duration will be computed from self-reported bed and wake up times using sleep logs and measured using an Actiwatch.
Sleep Quality | Total of 2 weeks between Visit 1 and 3
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index and Insomnia Severity Index
Light Exposure | Total of 2 weeks between Visit 1 and 3
  Measured using Actiwatch
Total Energy Intake | Total of 2 weeks between Visit 1 and 3
  Total energy intake in kcal/day will be computed from 14-day 24-hr dietary recalls
Dietary Composition | Total of 2 weeks between Visit 1 and 3
  Macronutrient and micronutrient intake will be computed from 14-days of self-reported 24-hr dietary recalls
Dietary Intake Timing | Total of 2 weeks between Visit 1 and 3
  Food timing will be self-reported and averaged across 14-days of 24-hr dietary recalls
Physical Activity | Baseline
  Assessed using the International Physical Activity Questionnaire (IPAQ)
Chronotype | Baseline
  Assessed using the Morningness-Eveningness Questionnaire (MEQ)
Emotional Eating Behavior | Baseline
  Assessed using the Emotional Eating Questionnaire (EEQ)
Depression | Baseline
  Assessed using the Patient Health Questionnaire (PHQ-8)

CONTACTS AND LOCATIONS:
Overall Officials: Richa Saxena, PhD, Principal Investigator — Massachusetts General Hospital; Frank AJL Scheer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Recruitment Website — https://clinicaltrials.partners.org/study/shiftstudy